CLINICAL TRIAL: NCT05845034
Title: A New Theory of Electrophysiological Mechanism of Atrial Fibrillation and Catheter Ablation Therapy for Atrial Fibrillation
Brief Title: A New Theory of Electrophysiological Mechanism of Atrial Fibrillation
Acronym: ANTEMAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, mingli Zhou, Principal Investigator, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASE2022
Record Dates: First submitted 2023-04-01; First posted 2023-05-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With additional SPEs ablation (Experimental): Patients who undergo PVI + SPEs ablation using ThermoCool SmartTouch catheter.
  Interventions: Procedure: PVI + SPEs ablation
- Control Group (Active Comparator): Patients who undergo PVI alone using ThermoCool SmartTouch catheter.
  Interventions: Procedure: PVI ablation

INTERVENTIONS:
Procedure: PVI + SPEs ablation — electrophysiology substrate mapping is the critical difference between both groups.
  Arms: With additional SPEs ablation
Procedure: PVI ablation — electrophysiology substrate mapping is the critical difference between both groups.
  Arms: Control Group

SUMMARY:
The electrophysiological mechanisms of atrial fibrillation remain disagreements. The goal of this clinical trail is to propose a new electrophysiological mechanism hypothesis of atrial fibrillation（AF）,meanwhile, the investigators sought to test the hypothesis that the superposition electrograms (SPEs) recorded during atrial fibrillation could be used as target sites for catheter ablation of atrial fibrillation.

DETAILED DESCRIPTION:
Catheter ablation for atrial fibrillation is a promising therapy, whose success is limited in part by uncertainty in the electrophysiological mechanisms of AF. The investigators recruited 100 subjects including paroxysmal(40%) and persistent (60%) AF. Cases were prospectively treated, in a 2-arm 1:1 design, by ablation SPEs followed by pulmonary vein isolation(PVI) ablation (n=50), or pulmonary vein isolation alone (n =50).

All procedures are guided by CARTO (Biosense Webster) electroanatomic mapping system and ablation is performed using open irrigated catheters with contact force (CF) sensing (Thermocool SmartTouch, Biosense Webster). Study Group underwent electroanatomic mapping during AF. Using CARTO to identify areas associated with SPEs. Radiofrequency ablation of the area with SPEs was performed, aiming to eliminate SPEs and convert to sinus rhythm or atrial tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a first-time ablation procedure for AF
* Paroxysmal AF will be defined as a sustained episode lasting > 7 days; Persistent AF will be defined as a sustained episode lasting > 7 days and less than 1 years; Long-lasting persistent AF will be more than 1 year and less than 5 years.
* Patients must be willing and able to comply with all peri-ablation and follow-up requirements.
* Patients with atrial fibrillation will to accept the procedure of ablation.
* Patients signed the written informed consent for the study.
* Patients can endure the required follow up.

Exclusion Criteria:

* Patients with contraindications to systemic anticoagulation with heparin or a direct thrombin inhibitor.
* Patients with thromboembolus in left atrial appendage.
* Patients with left atrial size ≥ 55 mm (2D echocardiography, parasternal long-axis view).
* Patients allergic for contrast or iodine.
* Patients with the serum creatinine（SCr） >3.5mg/dl
* Patients with life expectancy < 12 months
* Patients who are in the period of pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF during follow-up | one year
  At the one-year follow-up，AF occurring in the first 3 months after the ablation (blanking period) were censored.Beyond this, any AF episode that lasted for more than 30 seconds was categorized as a recurrence.

SECONDARY OUTCOMES:
Acute success rate of AF termination during ablation procedure | one year
  Conversion of AF to normal sinus rhythm or atrial tachyarrhythmias during ablation procedure.
Complications | one year
  Serious adverse events included death, pericardial tamponade , cerebrovascular events, significant PV stenosis , left atrial-esophageal fistula.
freedom from documented AF/AT episode | one year
  freedom from any documented AF/AT episode lasting > 30 s after the blanking period without anti-arrhythmic drugs during the 12-month follow-up after a single procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mingli Zhou, M.D., Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Result] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410
- [Result] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076